CLINICAL TRIAL: NCT00832065
Title: Sexual Dysfunction And Hypotestosteronemia In Patients With Obstructive Sleep Apnea Syndrome And Its Effects With CPAP Therapy
Brief Title: Sexual Dysfunction And Hypotestosteronemia In Patients With Obstructive Sleep Apnea Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled in study
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-066
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea; Hypotestosteronism
Keywords: Sleep Apnea Syndrome; Sleep Apnea; CPAP; Low testosterone; Sexual Dysfunction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients With Sleep Apnea and Low Testosterone: Adult male patients between 18-70 years of age with nely diagnosed OSAS documented by all night polysomnography(PSG)

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS)is a common disease and is suspected to be associated with sexual dysfunction. Our purpose is to sudy the effect of CPAP (Continuous Positive Airway Pressure) treatment on patients' sexual dysfunction by measuring testosterone levels before and after CPAP treatments.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea Syndrome(OSAS) is a highly prevalent disease in the population, affecting at least 4% of males and to a lesser extent females, yet it is currently under diagnosed. OSAS is associated with various disorders including cardiovascular disease, insulin resistance, diabetes mellitus, fatigue and erectile dysfunction. Currently the standard treatment for OSAS is Continuous Positive Airway Pressure(CPAP).

Low testosterone levels are present in some patients with OSAS leading to erectile dysfunction. However, the true prevalence of low testosterone levels and its correlation with sexual health is poorly understood and undefined. Prior data suggest treating these patients with CPAP therapy, usually increases testosterone levels, but unclear if this makes any meaningful difference in patient outcome, that is improvement in libido and sexual function.

There are several postulations to the pathophysiology of low testosterone levels in patients with OSAS. CRP(C-reactive protein), a strong marker of inflammation was shown to be elevated in patients with OSAS. The association between elevated CRP and low testosterone level would support the notion that inflammation plays a primary role in sexual dysfunction in patients with OSAS.

The objective of this study is to identify correlation between low free testosterone levels, sexual dysfunction and Obstructive Sleep Apnea before and after treatment with CPAP. Evaluate the role of CRP and inflammation secondary to OSAS in the pathogenesis of sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult males ages 18-70 with newly diagnosed OSAS documented by all-night polysomnography (PSG)

Exclusion Criteria:

* Currently on testosterone replacement therapy
* Prior known cause of erectile dysfunction
* Patients with prior treatment of erectile dysfunction
* Co-morbid conditions like diabetes, hypertension, as well as patient medications, will be recorded, and will not be part of the exclusion criteria

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the departments of Pulmonary and Critical Care and Endocrinology Lahey Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Correlation between low free testosterone levels, sexual dysfunction and Obstructive Sleep Apnea before and after treatment with CPAP. Free testosterone levels and its affect with CPAP treatment | 3 months

SECONDARY OUTCOMES:
Sexual Function Assessments. Confirmation of a link between OSAS, elevated CRP levels, and low testosterone. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Akmal Sarwar, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (2):
- United States (2):
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Lahey Clinic Northshore, Peabody, Massachusetts

REFERENCES:
- [Background] Karacan I, Karatas M. Erectile dysfunction in sleep apnea and response to CPAP. J Sex Marital Ther. 1995 Winter;21(4):239-47. doi: 10.1080/00926239508414643. PMID 8789505
- [Background] Bratel T, Wennlund A, Carlstrom K. Pituitary reactivity, androgens and catecholamines in obstructive sleep apnoea. Effects of continuous positive airway pressure treatment (CPAP). Respir Med. 1999 Jan;93(1):1-7. doi: 10.1016/s0954-6111(99)90068-9. PMID 10464840
- [Background] Grunstein RR, Handelsman DJ, Lawrence SJ, Blackwell C, Caterson ID, Sullivan CE. Neuroendocrine dysfunction in sleep apnea: reversal by continuous positive airways pressure therapy. J Clin Endocrinol Metab. 1989 Feb;68(2):352-8. doi: 10.1210/jcem-68-2-352. PMID 2493027
- [Background] Goncalves MA, Guilleminault C, Ramos E, Palha A, Paiva T. Erectile dysfunction, obstructive sleep apnea syndrome and nasal CPAP treatment. Sleep Med. 2005 Jul;6(4):333-9. doi: 10.1016/j.sleep.2005.03.001. PMID 15946896
- [Background] Hoekema A, Stel AL, Stegenga B, van der Hoeven JH, Wijkstra PJ, van Driel MF, de Bont LG. Sexual function and obstructive sleep apnea-hypopnea: a randomized clinical trial evaluating the effects of oral-appliance and continuous positive airway pressure therapy. J Sex Med. 2007 Jul;4(4 Pt 2):1153-62. doi: 10.1111/j.1743-6109.2006.00341.x. Epub 2006 Nov 1. PMID 17081222
- [Background] Luboshitzky R, Lavie L, Shen-Orr Z, Lavie P. Pituitary-gonadal function in men with obstructive sleep apnea. The effect of continuous positive airways pressure treatment. Neuro Endocrinol Lett. 2003 Dec;24(6):463-7. PMID 15073577